CLINICAL TRIAL: NCT06581978
Title: Early Warning and Intervention Mechanism of Foot Health Risk in Children and Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2024-278
Record Dates: First submitted 2024-08-25; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Flexible Flatfoot
Keywords: Children; Flatfoot; Traditional Chinese medical exercises training; Wearable sensors; Whole body vibration
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole-Body Vibration Intervention Group (Experimental): Enrolled children will be trained at home using a vertical rhythm device under the guidance of researchers and parental supervision. WBV training lasted for four weeks, five days a week, 15 minutes a day, each movement lasted for 30 seconds, and 30 seconds of rest between groups.
  Interventions: Procedure: Exercise Intervention Group
- Control Group (No Intervention): Children were instructed to rest and not participate in physical activity
- Traditional Chinese medical exercises training Intervention Group (Experimental): The enrolled children will be supervised by their parents and follow the teaching of the self-developed APP for Yi Jin Jing exercises. The training lasts for 4 weeks, 5 days a week, 15 minutes a day, 12 movements in total, each movement is 1 minute, and the rest between groups is 15 seconds.
  Interventions: Procedure: Whole-Body Vibration Intervention

INTERVENTIONS:
Procedure: Whole-Body Vibration Intervention — Whole-Body Vibration Intervention
  Arms: Traditional Chinese medical exercises training Intervention Group
Procedure: Exercise Intervention Group — Traditional Chinese medical exercises training
  Arms: Whole-Body Vibration Intervention Group

SUMMARY:
This clinical study was a prospective intervention study. The growth and development parameters and kinematic parameters of 120 children were planned to be collected for an observational study, and then the sensors were used to collect long-term gait data for 4 weeks and record the occurrence of foot pain. Children were assigned to the observation group, exercises intervention group, or WBV vertical rhythm intervention group according to their wishes. After 4 weeks of intervention, the dynamic and static foot posture differences between the intervention group and the observation group were analyzed and compared.

DETAILED DESCRIPTION:
This clinical study plan to recruit 120 subjects aged 6-18 years to collect the following parameters:

1. Three-dimensional shape of foot: The three-dimensional shape parameters of foot are obtained by 3D morphometric scanner, which is harmless to human body and has no radiation. The subjects stand barefoot on a 3D morphometric scanner and test their left and right feet respectively.
2. Static foot posture: foot Posture Index-6, foot X-ray bearing position.
3. Bone age analysis: Bone age is measured by using the stereotype protected mobile wrist with microradiation amount.
4. Bone mineral density analysis: calcaneal bone mineral density is measured by musculoskeletal ultrasound.
5. Genome grouping: Children's saliva is collected for whole genome analysis.
6. Body fat analysis: Bioresistive method was used to evaluate body fat ratio.
7. TCM physique assessment: Classification and Identification of TCM physique of Children in Guangdong Region by TCM Physique Scale combined with tongue image analysis (T/GDACM 0112 -- 2022).
8. Passive optical motion capture system, plantar pressure system and surface EMG system are used to collect kinematic parameters.

A wearable sensor is used to collect gait data for more than 8 hours per day for 4 weeks, and all enrolled children wear the wearable sensor in their daily lives. The obtained data is uploaded to the cloud server through the mobile application, and the data is uploaded through the APP to achieve remote monitoring and daily event recording. When the subject has a foot pain event, it should be reported to the researchers through the APP in time. After determining the foot pain based on the VAS score, the foot pain subjects will be divided into the observation group, the exercise intervention group and the WBV vertical rhythm intervention group according to their willingness.

The children in the observation group followed the doctor's advice to rest and did not participate in sports activities. The children in the intervention group were followed up by the researchers to implement the WBV vertical rhythm or exercise training program. The follow-up time was once a week and the training lasted for 4 weeks. The self-developed APP was used for researchers to remotely monitor and guide children's training movements and track training progress. The device uses a Huawei S-TAG anklet that matches HarmonyOS 2+/Android 6.0+/iOS 9.0+. IP68 (GB/T 4208-2017), waterproof grade 50 meters; Bluetooth: BT 5.0 to transmit data; Running scenario battery life: running 1 hour a day, running 5 days a week, stationary placement when not in use, battery life of 30 days.

1. WBV vertical rhythm training standard procedure: Enrolled children will be trained at home using vertical rhythm equipment under the guidance of researchers and parental supervision. WBV training lasted for four weeks, five days a week, 15 minutes a day, each movement lasted for 30 seconds, and 30 seconds of rest between groups.
2. Standard process of TCM exercise training: The enrolled children will be supervised by their parents and follow the teaching of the self-developed APP for exercise training. The Yi Jin Jing training lasts for 4 weeks, 5 days a week, 15 minutes a day, 12 movements in total, each movement is 1 minute, and the rest between groups is 15 seconds. Improvement in static and dynamic foot posture is assessed at the end of the 4-week training period.

ELIGIBILITY:
Inclusion Criteria:

1. They agreed to participate in the study, and their legal representatives voluntarily signed an informed consent form
2. 6-18 years old typical development of children and adolescents, gender not limited

Exclusion Criteria:

1. In addition to the flat feet, there are other effects foot posture or spinal congenital malformation of the lower limbs
2. At the investigator's discretion, he was not considered to be suitable to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Static foot posture | Baseline , pre-intervention and immediately after the intervention
  Static foot posture is evaluated using 3D morphometric scanner, X-ray, and Foot Posture Index-6
Motional foot posture | Baseline , pre-intervention and immediately after the intervention
  Motional foot posture is evaluated using Passive optical motion capture, and wearable sensors

SECONDARY OUTCOMES:
Foot pain events | Baseline , pre-intervention
  Visual Analogue Scale (VAS) is used to evaluate foot pain, which asks patients to rate their pain level on a scale of 0 to 10 (0 = no pain; 10 = "worst pain ever"). On the VAS scale, patients draw a hash mark representing their pain level on an unmarked 10-cm line, with the left side marked as "no pain" and the right side marked as "unbearable pain".
Bone maturity | Baseline , pre-intervention
  Bone age taken by dual energy X ray bone age instrument, the equipment radiation is extremely low, the equivalent of flying two minutes, or about 20 minutes of walking in the sunshine, won't cause harm to human body. Bone mineral density (BMD) was measured by ultrasound bone densitometer, which can be used to measure the BMD of calcaneus in children without radiation and trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

DOCUMENTS (2):
  • Study Protocol (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT06581978/Prot_000.pdf
  • Informed Consent Form (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT06581978/ICF_001.pdf